CLINICAL TRIAL: NCT05047237
Title: eFIcacious-Diabetes Care: a Pilot Study of a Pharmacist-Led Optimization Intervention to Achieve Guideline-based Care for Frail Older Adults
Brief Title: Electronic Frailty Index (eFI)Cacious-Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00076190
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-09

CONDITIONS: Diabetes; Type2 Diabetes
Keywords: HbA1c; diabetes care; diabetes type 2; Guideline-Based Care; Pharmacist-Led Optimization
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Subjects in this arm will receive standard of care treatment with no intervention. They will receive month 6 follow up.
- Active Decliners (No Intervention): Subjects who decline intervention. Standard of care treatment with month 6 follow up.
- Active Intervention (Experimental): Subjects are mailed Information about Type 2 Diabetes Mellitus (T2DM) Guidelines and Appointment Information (Face to face [F2F] or Telehealth). They attend up to 3 pharmacist visits, depending on if they reach target glucose levels. And they attend interviews. They also have month 6 follow up.
  Interventions: Behavioral: Pharmacist-Led Optimization Intervention

INTERVENTIONS:
Behavioral: Pharmacist-Led Optimization Intervention — Educational information mailed to participants and up to three pharmacist visits.
  Arms: Active Intervention

SUMMARY:
The purpose of this research is to explore whether a pharmacist-led diabetes management program can help optimize diabetes care for older adults. Participation in this study will involve meeting with a pharmacist who works with subjects' doctors, getting some routine bloodwork typical for people with diabetes, and potentially adjusting the subject's diabetes medications to reach American Diabetes Association guidelines. This study aims to bring older adults with diabetes whose measurements and medications are different from the guidelines of the American Diabetes Association into guidelines-based ranges.

DETAILED DESCRIPTION:
This study is a pragmatic pilot study assessing the feasibility and acceptability, and preliminary impact of a pharmacist-led care pathway to align patient care with guidelines for type 2 diabetes mellitus (T2DM) management in frail older adults, leveraging existing resources and pathways of care led by Clinical Prescribing Pharmacists. Eligible participants will be identified from the Electronic Health Record (EHR). Research staff will then approach the primary care physicians for identified patients to confirm that patients are appropriate for the intervention, as determined by the primary care physician (PCP). Patients will then be contacted both by letter and phone call, and invited to participate in the pharmacist-led pathway. Telephonic informed consent will be obtained. Outcomes for all participants will be accessed passively via the EHR. The study team hypothesizes that patients who go through the pharmacist-led primary care intervention will be more likely to have guideline-concordant medical therapy as compared with an EHR-based control group. Also, the study team believes that the intervention will reach at least 50% of those referred by their physicians to participate, the median number of outpatient visits will be three or less, and that the intervention will require a total of <3 hours for pharmacists and patients across the 3-month intervention period. In addition, the study team expects patients, physicians, and pharmacists will report the intervention is feasible, acceptable, appropriate, and high-value. Lastly, the study team believes that the intervention group will have a lower mortality than the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Attributed to a Atrium Health Wake Forest Baptist-affiliated Accountable Care Organization
* At least 2 consecutive International Classification of Diseases 10th Revision (ICD-10) codes for type two diabetes mellitus in the prior 2 years
* Has a calculable Electronic Frailty Index (eFI) score >0.21
* A glycosylated hemoglobin (HbA1c) value <7.5% in the prior 2 years
* Currently taking a sulfonylurea or insulin for Type 2 Diabetes Mellitus (T2DM)

Exclusion Criteria:

* Moderate to severe hearing loss (due to phone interventions)
* Diagnosed Alzheimer's disease or related dementia (unable to participate)
* Non-English speaking (not all pharmacists speak a second language; subtleties may not be conveyed effectively)
* No phone number available for patient (follow up contacts will be by telehealth or phone

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who Achieve Glycosylated Hemoglobin (HbA1c) values | Month 6
  Proportion of subjects who achieve target value of HbA1c >7.5%
Change in HbA1c | From Baseline through Month 6
Random Glucose Measurements | From Baseline through Month 12
  The study team will track any glucose measurements obtained between initial enrollment and 6-12 months follow up after completion of the intervention, up until a total of 12 months after initial enrollment. This will be reported as a glucose trajectory.
Estimated Change in Out-of-Pocket Costs | From Baseline through Month 6
  Change in diabetes medication cost
Point estimates of Feasibility Measures: Participation/Reach | Month 6
  The proportion of those referred who chose to participate
Point estimates of Feasibility Measures: Number Contacted/Reach | Month 6
  Total number of subjects contacted
Point estimates of Feasibility Measures: Number at Risk/Reach | Month 6
  Total number of patients who meet inclusion/exclusion criteria at each site
Feasibility Measures: Effort Required to Enroll-Number Calls | Month 6
  Number of calls to enroll
Feasibility Measures: Effort Required to Enroll-Average Call Duration | Month 6
  Duration of calls to enroll in minutes.
Point estimates of Feasibility Measure-Number of Visits | Month 12
  Mean and median number of visits with the pharmacist before glucose levels are met.
Point estimates of Feasibility Measures: Time | Month 12
  Time until achieved medication goal per patient will be reported. An achieved medication goal is the following: HbA1c <8 while taking no sulfonylurea or insulin, or HbA1c between 7.5-8 on sulfonylurea or insulin (these would both meet guidelines-based care.

SECONDARY OUTCOMES:
Rate of Emergency Department Visits and Hospitalizations | Baseline through Month 18
  Using EHR and Patient Ping, the number of contacts with the Emergency Department (ED) and hospitals (composite)
Number of Hypoglycemic Events Requiring Medical Assistance | Time Frame: Baseline through Month 18
  Events defined as per action to control cardiovascular risk in diabetes (ACCORD) trial, as hypoglycemic episodes requiring hospitalization or care in an emergency department.
Number of Injurious Falls | Baseline through Month 18
  Identified by International Classification of Diseases-10th Revision (ICD-10) diagnostic codes; defined as per systolic blood pressure intervention trial (SPRINT) as falls requiring hospitalization or care in an emergency department.
Mortality | Baseline through Month 18
  Number of people who die as found in EHR and North Carolina (NC) death registry
Implementation Metric--Feasibility | Baseline through Month 18
  Feasibility (FIM): This is a questionnaire that helps determine feasibility of the intervention. Score ranges from 4-20, with a higher score meaning the participant feels the intervention is more feasible.
Implementation Metric-- Acceptability | Baseline through Month 18
  This is a questionnaire that helps determine acceptability of the intervention. Score ranges from 4-20, with a higher score meaning the participant feels the intervention is more acceptable.
Implementation Metric-- Appropriateness | Baseline through Month 18
  This is a questionnaire that helps determine appropriateness of the intervention. Score ranges from 4-20, with a higher score meaning the participant feels the intervention is more appropriate.
Implementation Metric- Value | Baseline through Month 18
  Three questions will be coded and analyzed through qualitative analysis. The study team will code comments by hand using content analysis and grounded theory.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E. Callahan, MD, Principal Investigator — Atrium Health Wake Forest Baptist Health
Locations (1):
- Atrium Health Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study, "eFIcacious-Diabetes Care: a Pilot Study of a Pharmacist-Led Optimization Intervention to Achieve Guideline-based Care for Frail Older Adults" agrees to share study data that fulfill the International Committee of Medical Journal Editors (ICMJE) requirements starting after the first 3 months after our study has started and five years after our first article publication. We agree to provide data to researchers who can provide our lab with a methodologically sound proposal, and who need our data to help achieve aims outlined in their proposal. The study's data will be comprised of individual participant data that underlie the results reported in our publication. Participant data will be deidentified and can be used in text, tables, figures, and appendices, after approval from the study's primary investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 mos and ending 5 years following article publication
Access Criteria: The requests must include a proposal with clear aims as to why and how the data will be used. If proposal is approved, a data access agreement will need to be signed and will only be accessible for a 5-year period. All requests to gain access to the data will need to be sent to the study's PI, Kathryn Callahan, MD, MS, (kecallah@wakehealth.edu).

DOCUMENTS (1):
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT05047237/ICF_000.pdf